CLINICAL TRIAL: NCT02446483
Title: Comparative Randomized, Single Dose, Two-way Crossover Open-label Study to Determine the Bioequivalence of Rabeprazole From Idiazole 20mg DR Tabs (GSK, Egypt)and PARIET 20 mg DR Tabs (JANSSEN, EGYPT) After a Single Oral Dose Administration of Each to Healthy Adults Under Fasting Conditions
Brief Title: A Bioequivalence Study of Idiazole 20mg DR Tabs and PARIET® 20 mg DR Tabs After a Single Oral Dose Administration Under Fasting Conditions in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201527
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Gastrointestinal Diseases
Keywords: Idiazole 20mg; PARIET 20 mg; Rabeprazole; bioequivalence
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Thirty subjects will receive a single oral dose of idiazole 20mg DR tabs under fasting condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of PARIET 20 mg DR tabs under fasting condition in treatment period 2.
  Interventions: Drug: Idiazole 20mg DR tabs; Drug: PARIET 20 mg DR tabs
- Group B (Experimental): Thirty subjects will receive a single oral dose of PARIET 20 mg DR tabs under fasting condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of idiazole 20mg DR tabs under fasting condition in treatment period 2.
  Interventions: Drug: Idiazole 20mg DR tabs; Drug: PARIET 20 mg DR tabs

INTERVENTIONS:
Drug: Idiazole 20mg DR tabs — Delayed release tablets containing 20 mg of rabeprazole
Drug: PARIET 20 mg DR tabs — Orally administered, delayed-release, enteric-coated tablets containing 20 mg of rabeprazole sodium.

SUMMARY:
This is an open-label, randomized, single dose, two-sequence, two-period crossover study, separated by 7 days washout interval from the first study drug administration.

In this study, the bioavailability of Rabeprazole from Idiazole 20 milligram (mg) delayed release (DR) tablets and PARIET 20 mg DR tablets after a single oral dose administration of each to healthy adults under fasting conditions, will be investigated by determining the 90% confidence limits for the log-transformed ratio (Test product / Reference product) for the bioequivalence parameters. The influence of sequence, product and period effect will be tested by analysis of variance (ANOVA).

In this study a total of 60 subjects plus 1-4 additional subjects will be enrolled and split into two groups (Group A and B) of 30 each. For each subject, a total of 33 blood draws will be done and the volume of blood will not exceed 300 milliliters (mL) for the study.

PARIET is a registered trademark of EISAI Co. Limited.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, age 18 to 55 years, inclusive.
* Body weight within 10 percent of normal range according to the accepted normal values for body mass index (BMI).
* Medical demographics without evidence of clinically significant deviation from normal medical condition.
* Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
* Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

* Subjects with known allergy to the products tested.
* Subjects whose values of BMI were outside the accepted normal ranges.
* Female subjects who were pregnant, nursing or taking birth control pills.
* Medical demographics with evidence of clinically significant deviation from normal medical condition.
* Results of laboratory tests which are clinically significant.
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
* Subject is on a special diet (for example subject is vegetarian).
* Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
* Subject has a history of severe diseases which have direct impact on the study. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
* Subject intends to be hospitalized within 6 weeks after first study drug administration.
* Subjects who, through completion of this study, would have donated more than 500 mL of blood in 7 days, or 750 mL of blood in 30 days, 1000 mL in 90 days, 1250 mL in 120 days, 1500 mL in 180 days, 2000 mL in 270 days, 2500 mL of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2014-03-26 (Actual); Study Completion 2014-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201527 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201527 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201527 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201527 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201527 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 60 adult healthy male and female participants, aged 18 to 55 years, at a single site of Egypt from 30 January 2014 to 27 October 2014. During each study period participants received test (treatment A- rabeprazole tablet) and reference (treatment B-rabeprazole tablet) products.
Pre-assignment Details: Out of 64 participant screened, one participant was excluded because of significant variation in laboratory results and three participant withdrew the consent, remaining 60 were included in period I.
Groups:
- Treatment A-rabeprazole 20mg,Then Treatment B-rabeprazole 20mg: Participants received one tablet of treatment A (rabeprazole 20 milligram [mg] enteric coated tablet) given with 240 milliliter (mL) water according to a plan of randomization. Water was at room temperature and measured with a 250 mL cylinder. After a washout period of 7 days, participants then received one tablet of treatment B (rabeprazole 20 mg gastro-resistant tablet) given with 240 mL water. Participants were admitted the night before study drug administration, supervised for at least 10 hours (h) of overnight fasting, and confined until collecting 12 h blood sample during study drug administration of each period. The study drug administration took place between 10:00 ante meridiem (am) and 10:51 am on Day 1 of each study period.
- Treatment B-rabeprazole 20mg,Then Treatment A-rabeprazole 20mg: Participants received one tablet of treatment B (rabeprazole 20 mg gastro-resistant tablet) given with 240 mL water according to a plan of randomization. Water was at room temperature and measured with a 250 mL cylinder. After a washout period of 7 days, participants then received one tablet of treatment A (rabeprazole 20 mg enteric coated tablet) given with 240 mL water. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 12 h blood sample during study drug administration of each period. The study drug administration took place between 10:00 am and 10:51 am on Day 1 of each study period.
Period: Period 1: Intervention Period 1
Arm/Group | Treatment A-rabeprazole 20mg,Then Treatment B-rabeprazole 20mg | Treatment B-rabeprazole 20mg,Then Treatment A-rabeprazole 20mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 2: Washout Period (7 Days)
Arm/Group | Treatment A-rabeprazole 20mg,Then Treatment B-rabeprazole 20mg | Treatment B-rabeprazole 20mg,Then Treatment A-rabeprazole 20mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 3: Intervention Period 2
Arm/Group | Treatment A-rabeprazole 20mg,Then Treatment B-rabeprazole 20mg | Treatment B-rabeprazole 20mg,Then Treatment A-rabeprazole 20mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment A-rabeprazole 20 mg + Treatment B-rabeprazole 20 mg: In each period of the study, participants received one tablet of treatment A (rabeprazole 20 mg enteric coated tablet) or treatment B (rabeprazole 20 mg gastro-resistant tablet), given with 240 mL water according to a plan of randomization. Water was at room temperature and measured with a 250 mL cylinder. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 12 h blood sample during study drug administration of each period. The study drug administration took place between 10:00 am and 10:51 am on Day 1 of each study period. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Treatment A-rabeprazole 20 mg + Treatment B-rabeprazole 20 mg
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.72 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Region of Enrollment [Number; unit: Participants]
  Egypt | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximal Measured Plasma Concentration (Cmax) After a Single Dose
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at indicated time points of each treatment period. Cmax was defined as maximal measured plasma concentration over the time span specified. Values were reported as Least Squares Geometric Means with respective Geometric Coefficient of Variation (% CV).
Time Frame: Pre-dose (0.00) and 0.50, 1.00, 1.50, 2.00, 2.33, 2.66, 3.00, 3.33, 3.66, 4.00, 4.33, 4.66, 5.00, 5.33, 5.66, 6.00, 8.00, 12.00 and 14.00 h post-dose in each treatment period.
Population: All subject population comprised of all participants who were crossed over and completed the balance design, were included in the calculation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per mL (ng/mL)
Groups:
- Treatment A- Rabeprazole 20 mg: In each period of the study, participants received one tablet of treatment A (rabeprazole 2 mg enteric coated tablet) with 240 mL of water either in sequence of treatment AB or treatment BA as per the randomization. Water was at room temperature and measured with a 250 mL cylinder. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 12 h blood sample during study drug administration of each period. The study drug administration took place between 10:00 am and 10:51 am on Day 1 of each study period. The two treatment periods were separated by a washout period of 7 days.
- Treatment B- Rabeprazole 20 mg: In each period of the study, participants received one tablet of treatment B (rabeprazole 20 mg gastro-resistant tablet) with 240 mL of water either in sequence of treatment AB or treatment BA as per the randomization. Water was at room temperature and measured with a 250 mL cylinder. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 12 h blood sample during study drug administration of each period. The study drug administration took place between 10:00 am and 10:51 am on Day 1 of each study period. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Treatment A- Rabeprazole 20 mg | Treatment B- Rabeprazole 20 mg
Number analyzed (Participants) | 60 | 60
Nanogram per mL (ng/mL) | 543.78 (35.67) | 530.34 (32.98)
Statistical Analysis 1: Comparison: Treatment A- Rabeprazole 20 mg vs Treatment B- Rabeprazole 20 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence was established when 90% Confidence Interval falls within 80-125%; Point Estimate Percent = 101.32, 90% CI 2-sided [95.81 to 107.15]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) and Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-infinity)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. AUC0-t was calculated by the linear trapezoidal method. AUC0-infinity was calculated as the sum of the AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant, where first-order elimination or terminal rate constant was calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations. Values were reported as Least Squares Geometric Means with respective % CV.
Time Frame: as for outcome 1
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Treatment A- Rabeprazole 20 mg | Treatment B- Rabeprazole 20 mg
Number analyzed (Participants) | 60 | 60
ng.h/mL
  AUC0-t | 916.07 (43.30) | 922.52 (40.97)
  AUC0-infinity: number analyzed (Participants) | 56 | 57
  AUC0-infinity | 971.38 (41.98) | 959.78 (42.21)
Statistical Analysis 1: Comparison: Treatment A- Rabeprazole 20 mg vs Treatment B- Rabeprazole 20 mg; Comparison of T- rabeprazole 20 mg and R- rabeprazole 20 mg for AUC0-t; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; Point Estimate Percent = 98.71, 90% CI 2-sided [92.54 to 105.28]
Statistical Analysis 2: Comparison: Treatment A- Rabeprazole 20 mg vs Treatment B- Rabeprazole 20 mg; Comparison of Treatment A- rabeprazole 20 mg and Treatment B- rabeprazole 20 mg for AUC0-infinity; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; Point Estimate Percent = 98.05, 90% CI 2-sided [91.81 to 104.71]

3. Secondary Outcome: Time of the Maximum Plasma Concentration (T-max) and Terminal Half-life (T-half)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. If the maximum value occurs at more than one point T-max was defined as the first time point with this value. The elimination or terminal half-life was calculated by dividing 0.693 (natural logarithm of 2) with b obtained as the slope of the linear regression of the logarithmically transformed plasma concentrations versus time in the terminal period of the plasma curve.
Time Frame: as for outcome 1
Population: All Subject Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | Treatment A- Rabeprazole 20 mg | Treatment B- Rabeprazole 20 mg
Number analyzed (Participants) | 60 | 60
h
  Tmax | 2.66 [1.50 to 5.66] | 3.00 [1.50 to 8.00]
  T-half: number analyzed (Participants) | 56 | 57
  T-half | 2.79 [0.23 to 6.27] | 2.50 [0.70 to 5.73]
Statistical Analysis 1: Comparison: Treatment A- Rabeprazole 20 mg vs Treatment B- Rabeprazole 20 mg; Test type: Superiority or Other; p = 0.0029, Wilcoxon's Signed-Rank Test

4. Secondary Outcome: Apparent First-order Elimination or Terminal Rate Constant
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. Apparent first-order elimination or terminal rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: All subject population. Data is presented for the participants available at the time of assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | Treatment A- Rabeprazole 20 mg | Treatment B- Rabeprazole 20 mg
Number analyzed (Participants) | 56 | 57
Per hour | 0.35 (123.31) | 0.28 (46.12)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAE) were reported through out the study (up to 11 days)
Description: AE and SAE were reported in all subject population.
Arm/Group | Treatment A- Rabeprazole 20 mg | Treatment B- Rabeprazole 20 mg
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.